CLINICAL TRIAL: NCT07401329
Title: Early and Late Neutrophil CD64 and Monocyte HLA-DR as Biomarkers for Septic Shock
Status: Completed | Type: Observational
Sponsor: Pandit Bhagwat Dayal Sharma, PGIMS, Rohtak (Other)
Responsible Party: Principal Investigator, Aman Ahuja, Assistant Professor, Department of PCCM, Pandit Bhagwat Dayal Sharma, PGIMS, Rohtak
Other Study IDs: BREC/18/194
Record Dates: First submitted 2026-01-14; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Sepsis; Septic Shock
Keywords: HLADR; NCD64; sepsis; septic-shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic shock group
- Control group

SUMMARY:
Study Summary: Neutrophil CD64 & Monocyte HLA-DR in Septic Shock

What is studied?

Doctors looked at two blood markers:

* Neutrophil CD64 (nCD64): rises quickly when the body fights infection.
* Monocyte HLA-DR (mHLA-DR): falls when the immune system becomes weak or "paralyzed." They also calculated a Sepsis Index (ratio of nCD64 to HLA-DR) to see how these markers change in patients with septic shock.

Why is this important? Septic shock is a severe form of sepsis that can cause organ failure and death. Early detection and knowing which patients are at higher risk can guide treatment and improve survival.

How was it done?

* Blood samples were taken on Day 1 (early) and Day 8 (late).
* Results will be compared between survivors and non-survivors.
* 20 healthy people provided baseline values for comparison.

What does this mean? - Monitoring these markers over time (not just once) may helps doctors understand whether a patient's immune system is recovering or worsening.

Take-home message

For patients and families:

- Septic shock is serious, but doctors now have better tools to track how the body is responding.

DETAILED DESCRIPTION:
Detailed Protocol of the Study

1. Title Early and late neutrophil CD64 and monocyte HLA-DR as biomarkers for septic shock.
2. Study Design

   * Type: Prospective, single-center, observational cohort study.
   * Setting: Medical ICU of a tertiary care university teaching hospital in northern India.
   * Duration: January 2019 - December 2019.
   * Ethics Approval: Biomedical Research and Ethics Committee (BREC/18/194).
   * Guidelines: Conducted in adherence with STROBE reporting standards.
3. Objectives

   - Primary Objective: To evaluate neutrophil CD64 (nCD64), monocyte HLA-DR (mHLA-DR), and the Sepsis Index as prognostic markers in septic shock.
   * Secondary Objectives:
   * Compare biomarker levels between survivors and non-survivors.
   * Assess predictive accuracy of these markers for 28-day mortality using ROC analysis.
4. Study Population

   * Inclusion Criteria:
   * Age ≥18 years.
   * Diagnosis of septic shock according to prevailing Sepsis-3 criteria.
   * Written informed consent from patient or next of kin.
   * Exclusion Criteria:
   * Pregnant females.
   * Active malignancy.
   * Severe chronic liver disease.
   * Chronic kidney disease requiring maintenance hemodialysis.
   * Immunocompromised patients or those on immunomodulatory therapy prior to sepsis onset.
   * Non-bacterial sepsis (viral, fungal, tubercular).
5. Enrollment & Sample Size

   * Screened: 80 patients.
   * Excluded: 24 (per exclusion criteria).
   * Final cohort: 56 patients (37 survivors, 19 non-survivors).
   * Controls: 20 healthy volunteers for baseline biomarker values.
6. Data Collection

   * Demographics: Age, sex, residence, BMI, smoking status.
   * Clinical variables: Primary diagnosis, comorbidities, severity scores (qSOFA, SIRS, APACHE II), vital signs, organ dysfunction parameters (PaO₂/FiO₂, inotropic support, renal replacement therapy, GCS).
   * Laboratory parameters: CBC, renal/liver function tests, ABG, primary diagnosis details.
   * Outcome measures: ICU stay, ventilator days, 28-day mortality.
7. Biomarker Assessment

   * Markers:
   * Neutrophil CD64 (nCD64).
   * Monocyte HLA-DR (mHLA-DR).
   * Sepsis Index = nCD64 ÷ mHLA-DR.
   * Method: Flow cytometry (8-color FACS Canto II, BD Biosciences).
   * Units: Mean Fluorescence Intensity (MFI).
   * Time points:
   * Day 1 (admission).
   * Day 8 (follow-up).
8. Statistical Analysis

   * Software: SPSS v24 (IBM).
   * Descriptive statistics: Mean ± SD for normal data; median (IQR) for skewed data.
   * Comparisons:
   * Independent t-test for normal distribution.
   * Mann-Whitney U test for skewed data.
   * Predictive analysis: ROC curves for nCD64, HLA-DR, and Sepsis Index.
   * Significance threshold: p < 0.05 (two-sided).
9. Outcomes

   * Primary outcome: 28-day mortality.
   * Secondary outcomes: ICU stay duration, ventilator days, organ dysfunction severity.
10. Safety & Compliance

    * Biomedical waste: Managed per Biomedical Waste (Management and Handling) Rules.
    * Patient safety: Standard ICU protocols followed; no intervention beyond routine care.

ELIGIBILITY:
Inclusion Criteria: Patients were eligible if they met all of the following:

* Age ≥ 18 years.
* Diagnosis of septic shock according to prevailing Sepsis-3 criteria at the time of study.
* Admission to the medical ICU of the tertiary care teaching hospital.
* Written informed consent obtained from patient or next of kin.

Exclusion Criteria: Patients were excluded if they met any of the following:

* Pregnant females.
* Active malignancy (any known cancer diagnosis).
* Severe chronic liver disease.
* Chronic kidney disease requiring maintenance hemodialysis.
* Immunocompromised state, including:
* HIV/AIDS.
* Long-term corticosteroid therapy.
* Other immunosuppressive conditions.
* Prior immunomodulatory treatment before onset of sepsis (e.g., biologics, GM-CSF, interferons).
* Non-bacterial sepsis, including:
* Viral sepsis.
* Fungal sepsis.
* Tubercular sepsis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients aged over 18 years with a diagnosis of septic shock
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Measure the concentration of nCD64, mHLA-DR in mean fluorescence intensity (MFI) on day 1 and 8 | from day of enrollment to day 8
  * Sample Collection: Peripheral blood samples taken from patients with septic shock.
  * Technique: Flow cytometry using an 8-color FACS Canto II (BD Biosciences).
  * Units: Results expressed as Mean Fluorescence Intensity (MFI).
  * Calculation:
  * nCD64 measured directly on neutrophils.
  * mHLA-DR measured directly on monocytes.
To compare sepsis index on day 1 and day 8 | From day of enrollment to day 8
  Sepsis Index = nCD64 ÷ mHLA-DR.

SECONDARY OUTCOMES:
Compare the concentration of nCD64, mHLA-DR MFI between survivors and non-survivors. | from enrollment to day 28
  * Population: septic shock patients (survivors and non-survivors).
  * Time points: Day 1 (early) and Day 8 (late).
  * Markers: nCD64 (neutrophil CD64), mHLA-DR (monocyte HLA-DR)
  * Outcome: 28-day mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Dhruva Chaudhry, MBBS,MD,DM, Study Director — Pandit BD Sharma Postgraduate Institute of Medical Sciences
Locations (1):
- Pandit Bhagwat Dayal Sharma Postgraduate Institute of Medical Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Undecided